CLINICAL TRIAL: NCT05644483
Title: Effect of Remimazolam-remifentanil Versus Propofol-remifentanil Based General Anesthesia on Intraoperative Hemodynamic Stability in Prone Position for Major Spine Surgery: a Randomized Controlled Trial
Brief Title: Effect of Remimazolam and Propofol on Hemodynamic Stability in Prone Position
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical Assistant Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-1514
Record Dates: First submitted 2021-11-03; First posted 2022-12-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Hemodynamic Instability
Keywords: propofol; remimazolam
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- remimazolam group (Experimental): patients who receive remimazolam-remifentanil based total intravenous anesthesia
  Interventions: Drug: Remimazolam
- propofol group (Active Comparator): patients who receive propofol-remifentanil based total intravenous anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam: loading (6mg/kg/hr) + continuous infusion (1-2mg/kg/hr)
  Arms: remimazolam group
Drug: Propofol — Propofol: target controlled infusion: 2-3mcg/mL
  Arms: propofol group

SUMMARY:
Most of the major spinal surgeries are performed in the supine position, which causes a decrease in stroke volume and cardiac index, which leads to the occurrence of hypotension during surgery. Postoperative hypotension causes an imbalance in the supply and demand of oxygen, leading to postoperative myocardial infarction or acute renal damage, and may increase mortality one year after surgery. Propofol, which is most commonly used for total intravenous anesthesia, can further increase the incidence of hypotension during surgery. Therefore, there is a continuing demand for an anesthetic agent that is more hemodynamically stable. Remimazolam, an ultra-short acting benzodiazepine that has a similar structure to midazolam, but whose activity is terminated by esterase hydrolysis, is expected to have less hemodynamic effects than propofol. Therefore, the purpose of this study is to investigate the effect of general anesthesia using remimazolam and general anesthesia using propofol on hemodynamic safety during surgery in patients undergoing major spinal surgery in the supine position.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status: 1-3
* age: 19-80 years
* patients who are scheduled to undergo a major spine surgery in the prone position

Exclusion Criteria:

* patients who refuse to participate
* body mass index: <15kg/m2 or >35kg/m2
* patients with uncontrolled hypertension, hyperthyroidism, severe cardiac disease
* patients who are contraindicated to the use of remimazolam including severe hepatic disease, acute glaucoma, shock, acute alcohol intoxication
* allergic to propofol and midazolam
* patients who are judged unsuitable to participate in the study for other reasons by medical staffs

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
the number of hypotensive episode per patient | for one hour after turning the patients to the prone position
  SAP < baseline SBP * 80% or 90mmHg // MAP < baseline MAP * 80% or 65mmHg
the number of severe hypotensive episode per patient | for one hour after turning the patients to the prone position
  SAP < baseline SBP * 70% or 80mmHg // MAP < baseline MAP * 70% or 55mmHg

SECONDARY OUTCOMES:
cardiac index | for one hour after turning the patients to the prone position
  cardiac index from Flotrac
pleth variability index | for one hour after turning the patients to the prone position
  pleth variability index
heart rate | for one hour after turning the patients to the prone position
  heart rate from EKG
Total opioid consumption | for one hour after turning the patients to the prone position
  amount of total opioid administered
cardiac output | for one hour after turning the patients to the prone position
  cardiac output from Flotrac
stroke volume | for one hour after turning the patients to the prone position
  stroke volume from Flotrac
stroke volume variation | for one hour after turning the patients to the prone position
  stroke volume variation from Flotrac

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No